CLINICAL TRIAL: NCT02194452
Title: Efficacy of 68Ga-DOTATOC Positron Emission Tomography (PET) CT in Children and Young Adults With Brain Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sue O'Dorisio (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ride for Kids (Unknown)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Professor Pediatrics-HEM-Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201302711; P30CA086862 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Acoustic Schwannoma; Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Meningioma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Choroid Plexus Tumor; Adult Craniopharyngioma; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade I Meningioma; Adult Grade II Meningioma; Adult Medulloblastoma; Adult Meningeal Hemangiopericytoma; Adult Mixed Glioma; Adult Myxopapillary Ependymoma; Adult Oligodendroglioma; Adult Papillary Meningioma; Adult Pilocytic Astrocytoma; Adult Pineal Gland Astrocytoma; Adult Pineoblastoma; Adult Pineocytoma; Adult Subependymal Giant Cell Astrocytoma; Adult Subependymoma; Adult Supratentorial Primitive Neuroectodermal Tumor (PNET); Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Supratentorial Ependymoma; Meningeal Melanocytoma; Newly Diagnosed Childhood Ependymoma; Recurrent Adult Brain Tumor; Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Anaplastic Oligoastrocytoma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Diffuse Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Fibrillary Astrocytoma; Recurrent Childhood Gemistocytic Astrocytoma; Recurrent Childhood Giant Cell Glioblastoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Gliomatosis Cerebri; Recurrent Childhood Gliosarcoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Oligoastrocytoma; Recurrent Childhood Oligodendroglioma; Recurrent Childhood Pilocytic Astrocytoma; Recurrent Childhood Pilomyxoid Astrocytoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Pleomorphic Xanthoastrocytoma; Recurrent Childhood Protoplasmic Astrocytoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma; Recurrent Childhood Visual Pathway Glioma; Untreated Childhood Anaplastic Astrocytoma; Untreated Childhood Anaplastic Oligodendroglioma; Untreated Childhood Brain Stem Glioma; Untreated Childhood Cerebellar Astrocytoma; Untreated Childhood Cerebral Astrocytoma; Untreated Childhood Diffuse Astrocytoma; Untreated Childhood Fibrillary Astrocytoma; Untreated Childhood Gemistocytic Astrocytoma; Untreated Childhood Giant Cell Glioblastoma; Untreated Childhood Glioblastoma; Untreated Childhood Gliomatosis Cerebri; Untreated Childhood Gliosarcoma; Untreated Childhood Medulloblastoma; Untreated Childhood Oligoastrocytoma; Untreated Childhood Oligodendroglioma; Untreated Childhood Pilocytic Astrocytoma; Untreated Childhood Pilomyxoid Astrocytoma; Untreated Childhood Pineoblastoma; Untreated Childhood Pleomorphic Xanthoastrocytoma; Untreated Childhood Protoplasmic Astrocytoma; Untreated Childhood Subependymal Giant Cell Astrocytoma; Untreated Childhood Supratentorial Primitive Neuroectodermal Tumor; Untreated Childhood Visual Pathway and Hypothalamic Glioma; Untreated Childhood Visual Pathway Glioma
MeSH Terms: conditions — Neuroma, Acoustic; Astrocytoma; Ependymoma; Meningioma; Oligodendroglioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Glioma; Pinealoma; Glioma, Subependymal; Brain Neoplasms; Familial ependymoma; Neoplasms, Neuroepithelial; Optic Nerve Glioma | interventions — gallium Ga 68 dotatate; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (gallium Ga 68-edotreotide PET/CT) (Experimental): Patients undergo gallium Ga 68-edotreotide PET/CT at baseline and 1-30 days after surgery.
  Interventions: gallium Ga 68-edotreotide, positron emission tomography, computed tomography, laboratory biomarker analysis
  Interventions: Radiation: gallium Ga 68-edotreotide; Procedure: positron emission tomography; Procedure: computed tomography; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: gallium Ga 68-edotreotide — Undergo gallium Ga 68-edotreotide PET/CT
  Other Names: Ga-68 DOTA0-Tyr3-octreotide, Ga-68 DOTATOC
Procedure: positron emission tomography — Undergo gallium Ga 68-edotreotide PET/CT
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed
Procedure: computed tomography — Undergo gallium Ga 68-edotreotide PET/CT
  Other Names: tomography, computed
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies gallium Ga 68-edotreotide (68Ga-DOTATOC) positron emission tomography (PET)/computed tomography (CT) in finding brain tumors in younger patients. Diagnostic procedures, such as gallium Ga 68-edotreotide PET/CT imaging, may help find and diagnose brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if 68Ga-DOTATOC (gallium Ga 68-edotreotide) PET when combined with magnetic resonance imaging (MRI) will differentiate embryonal tumors such as medulloblastoma and supratentorial primitive neuroectodermal tumor (PNET) from the low and high grade gliomas.

II. To determine if 68Ga-DOTATOC PET will aid in the identification of residual tumor post operatively in those patients who were 68Ga-DOTATOC PET positive prior to surgery.

OUTLINE:

Patients undergo gallium Ga 68-edotreotide PET/CT at baseline and 1-30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with brain tumors will be eligible for this study
* Eligible subjects must be able and willing to undergo the procedures of the study
* Electronic version of pre-surgery MRI must be available for co-registration purposes
* Fresh frozen tumor, and/or paraffin block of biopsy or resected tumor is recommended, but not required to determine expression of somatostatin receptors in tumor by immunohistochemistry and/or quantitative polymerase chain reaction (qPCR)

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin of body that would preclude obtaining an MRI as part of the initial study evaluation
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons
* Presence of any additional medical condition such as inter-current illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance

Ages: 6 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in standardized uptake value (SUV) uptake after gallium Ga 68-edotreotide | Baseline up to 30 days
  The endpoint is a binary outcome (+ or -) of SUV uptake (after gallium Ga 68-edotreotide) and a binary outcome confirmed at biopsy (+ or -).
Proportion of discordance and concordance between gallium Ga 68-edotreotide and biopsy | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: M. Sue O'Dorisio, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States